CLINICAL TRIAL: NCT05439200
Title: Video Treatment for Amblyopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Eileen Birch, Senior Research Scientist, Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFSW113B; R01EY022313 (NIH)
Record Dates: First submitted 2022-06-17; First posted 2022-06-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asynchronous movies (Experimental): Asynchronous 3D movies
  Interventions: Device: Asynchronous 3D movies
- Standard-of-care patching with an adhesive patch (Active Comparator): Standard-of-care patching with an adhesive patch
  Interventions: Device: Patching

INTERVENTIONS:
Device: Asynchronous 3D movies — 3D movies streamed at home for viewing on a handheld lenticular 3D screen
  Arms: Asynchronous movies
Device: Patching — Adhesive patch to cover the fellow eye
  Arms: Standard-of-care patching with an adhesive patch

SUMMARY:
The purpose of this study is to determine whether viewing asynchronous movies leads to better visual outcomes in young children with amblyopia than standard-of-care occlusion therapy with an adhesive patch and whether this is associated with better adherence to treatment.

DETAILED DESCRIPTION:
This is a single-site randomized clinical trial to compare treatment of amblyopia by viewing asynchronous movies to standard-of-care occlusion therapy with an adhesive patch. Participants will be referred from local pediatric ophthalmologists. Following informed consent, children will complete baseline testing to confirm eligibility and provide pre-treatment measurements of visual acuity, suppression, stereoacuity, motor skills, self-perception, and quality of life. Eligible children will then be randomly allocated to either patch-free occlusion therapy or standard-of-care occlusion therapy with an adhesive patch.

Children will participate in their assigned occlusion therapy at home for 6 weeks (primary outcome). Adherence will be objectively monitored. Vision will be re-assessed at 2 and 4 weeks and all tests will be repeated at 6 weeks. The asynchronous movie group will have an option to continue for and additional 2 or 4 weeks (10 weeks total). The standard-of-care occlusion group will be offered the opportunity to use the movie treatment at the 6 week visit through 10 weeks. Children who choose to remain in the study beyond the 6 week primary outcome visit will have vision reassessed at 8 and 10 weeks.

The primary analysis will be a comparison of improvement in amblyopic eye visual acuity (baseline-6 weeks) between the movie group and the standard-of-care patching group. Secondary analyses will include comparisons of adherence to each treatment, comparison of the proportion of children in each group with visual acuity ≤0.1 logMAR (recovered) at 6 weeks and 95% CIs, comparisons of changes in extent of suppression, depth of suppression, stereoacuity, motor skills standard scores, self-perception scores, and PedEyeQ domain scores. Associations among hours of treatment, changes in visual acuity, suppression, and stereoacuity, will be explored and modeled for dose-response relationships. In exploratory analyses, we will examine whether there are additional improvements in visual acuity, suppression, or stereoacuity between 6 and 10 weeks for the movie group (8 and 10 weeks means and 95% CIs).

ELIGIBILITY:
Inclusion Criteria:

* aged 3-7 years
* male and female
* strabismic, anisometropic, or combined mechanism amblyopia (visual acuity 0.3-0.8 logMAR)
* interocular visual acuity difference ≥0.3 logMAR
* wearing glasses (if needed) for a minimum of 8 weeks with no change in visual acuity at 2 visits ≥4 weeks apart
* child's ophthalmologist and family willing to forgo standard patching treatment during the study

Exclusion Criteria:

* prematurity ≥8 wk
* coexisting ocular or systemic disease
* developmental delay
* strabismus >5 pd
* myopia > -3.00D

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in amblyopic eye visual acuity using a logMAR chart | 6 weeks
  change in amblyopic eye logMAR visual acuity relative to baseline

SECONDARY OUTCOMES:
Change in amblyopic eye visual acuity using a logMAR chart | 2, 4, 8, and 10 weeks
  change in amblyopic eye logMAR visual acuity relative to baseline at 2, 4, 8, and 10 weeks
Change in extent suppression assessed with the W4 test | 6 weeks
  change in log deg assessed with the W4 test relative to baseline
Change in stereoacuity assessed with the Randot Preschool Stereoacuity Test | 6 weeks
  change in log arcsec in stereoacuity assessed with the Randot Preschool Stereoacuity Test
Change in motor skills assessed with the Movement Assessment Battery for Children -2 | 6 weeks
  change in standard scores obtained with the Movement Assessment Battery for Children -2 (MABC-2; (normed and scaled 0-19, with 10 as an average score, 5-6 as "at risk", and <5 as "significant impairment")
Change in self perception assessed with the Pictorial Scale of Perceived Competence and Social Acceptance for Young Children | 6 weeks
  change in domain scores of the Pictorial Scale of Perceived Competence and Social Acceptance for Young Children (standard scores scaled to range from 0 to 100 for worst to best)
Change in quality of life assessed with the Pediatric Eye Questionnaire | 6 weeks
  change in domain scores of the Pediatric Eye Questionnaire (PedEyeQ; Rasch calibrated and scaled to score from 0 to 100 for worst to best)
Proportion of children who have recovered | 2, 4, 6, 8, and 10 weeks
  proportion of children who attain amblyopic eye visual acuity of at least 0.1 logMAR
Adherence to patching measured with a sensor and adherence to viewing videos measured with the streaming log data | 2,4, and 6 weeks
  cumulative hours of treatment with the patch objectively monitored temperature sensitive Theramon sensor or with movie viewing by monitoring the streaming logs
Change in depth of suppression assessed with the contrast balance index | 6 weeks
  change in contrast balance index (ratio of amblyopic eye to fellow eye contrast needed to overcome suppression

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Foundation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No